CLINICAL TRIAL: NCT01071564
Title: A Phase I Study of the Hedgehog Smoothened Antagonist GDC-0449 (NSC # 747691) Plus Pan-Notch Inhibitor RO4929097 (NSC # 749225) Administered in Patients With Advanced Breast Cancer
Brief Title: RO4929097 and Vismodegib in Treating Patients With Breast Cancer That is Metastatic or Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02064; NCI-2012-02064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000662081; 2009-099 (Other: Barbara Ann Karmanos Cancer Institute); 8420 (Other: CTEP); P30CA022453 (NIH); U01CA062487 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Pharmacogenomic Testing; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RO4929097 and vismodegib) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO on day 1 or days -2, -1, and 1 of course 1 and days 1-3 and 8-10 of course 2 and all subsequent courses. Patients also receive vismodegib PO QD beginning day 8 of course 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Pharmacological Study; Drug: Vismodegib

INTERVENTIONS:
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Pharmacological Study — Correlative studies
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase I trial studies the side effects and best dose of RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097) when given together with vismodegib in treating patients with breast cancer that is metastatic or cannot be removed by surgery. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as vismodegib, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving RO4929097 and vismodegib together may slow the growth of tumor cells and may be a more active treatment for advanced breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of continuous daily administration of 150 mg/day of GDC0449 (vismodegib) in combination with escalating doses of RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097) administered on a repeated schedule of days 1-3, 8-10 every 21 days (for a total of 6 days of RO4929097 administration per 21 day cycle) in patients with advanced breast cancer.

II. To determine the dose limiting toxicity (DLT) and identify the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) for this administration schedule.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics (PK) and pharmacogenetics (PG) of GDC0449 and RO4929097, each alone and in combination.

II. To attempt to evaluate select pharmacodynamic (PD) stem cell differentiation biomarkers in the hedgehog and notch signaling pathways (e.g. GLI family zinc finger [Gli]1/2/3, patched [Ptch] 1/2, hairy and enhancer of split 1, [Drosophila] [Hes1], huntingtin interacting protein 1 [Hip1], hairy/enhancer-of-split related with YRPW motif 1 [Hey1], Notch4, Jagged1, numb homolog [Drosophila] [numb], BMI1 polycomb ring finger oncogene [Bmi-1], cluster of differentiation [CD]44/CD24, aldehyde dehydrogenase [ALDH] proto-oncogene tyrosine-protein kinase [Src] family kinases) and the percentage of breast cancer stem cell (BCSC) in serial breast tumor biopsies before and after GDC0449 or RO4929097 alone and after 1 cycle of treatment with the combination of GDC0449 and RO4929097.

III. To determine tumor response in patients with measurable disease as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST).

IV. To perform molecular profiling of the tumor cell and BCSC populations before and after GDC0449 or RO4929097 alone and after 1 cycle of treatment with the combination of GDC0449 and RO4929097 at the MTD.

OUTLINE: This is a dose-escalation study of gamma-secretase/Notch signalling pathway inhibitor RO4929097.

Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) on day 1 or days -2, -1, and 1 of course 1 and days 1-3 and 8-10 of course 2 and all subsequent courses. Patients also receive vismodegib PO once daily (QD) beginning day 8 of course 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be women with histologically or cytologically confirmed locally advanced breast cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must be human epidermal growth factor receptor 2 (Her-2) non-expressing (if immunohistochemistry [IHC] 0 or 1+; fluorescent in situ [FISH] ratio less than 2; if IHC 2+, FISH ratio must be less than 2.0); once the MTD has been determined, the expansion phase will be limited to patients with estrogen receptor (ER), progesterone receptor (PR), and HER2 negative (i.e. "triple negative") disease; Her-2 will be assessed as above; ER and PR are considered negative if immunoperoxidase staining of tumor cell nuclei is < 5%
* Patients must have measurable disease per RECIST guidelines or evaluable (non-measurable) disease
* Patients MUST have tumor accessible and suitable for serial biopsy with 4-6 passes of a 16 or 18 gauge needle
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Prior therapy:

  * Patients must have failed at least 1 prior systemic therapy for metastatic or locally advanced breast cancer
  * IMPORTANT: Patients with chronic grade 1 or 2 toxicity may be eligible at the discretion of the Principal Investigator (e.g. grade 2 chemo-induced neuropathy); note that patients with ongoing alopecia of any grade will be eligible
  * Chemotherapy: prior chemotherapy is allowed; patients must not have received chemotherapy for 3 weeks prior to the initiation of study treatment and must have full recovery from any acute effects of any prior chemotherapy; patients must not have had nitrosoureas or mitomycin C for 6 weeks prior to the initiation of study treatment
  * Radiation: prior radiation therapy is allowed; patients must not have received minimal radiation therapy (=< 5% of their total marrow volume) within 3 weeks prior to the initiation of study treatment; otherwise, patients must not have received radiation therapy (> 5% of their total marrow volume) within 4 weeks prior to the initiation of study treatment; patients who have received prior radiation to 50% or more of their total marrow volume will be excluded
  * Other therapies: prior experimental (non-Food and Drug Administration [FDA] approved) therapies and immunotherapies are allowed; patients must not have received these therapies for 30 days or five half- lives of the drug prior to the initiation of study treatment and must have full recovery from any acute effects of these therapies; patients who have prior treatment with either a gamma-secretase or hedgehog inhibitor will be excluded from participating in this study
  * Patients must not have received allogeneic stem cell transplant
* Patients must not have co-morbid condition(s) that, at the opinion of the investigator, prevent safe treatment
* Patients must not have active infection or fever > 38.5 degree Celsius (C)
* Patients must not be human immunodeficiency virus (HIV)+, hepatitis B+ or hepatitis C+ (active or previous treatment)
* All patients must provide archival tissue block or paraffin sample from archival tissue block (approximately 10 sections) for use in pharmacodynamic and pharmacogenomics correlative studies
* Patients must agree to undergo a total of three serial biopsies for research purposes
* Patients with brain metastases will be eligible if condition is treated and stable for >= 1 month
* Patients must have a life expectancy of greater than 12 weeks
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets (PLT) >= 100,000/mcL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN); if liver metastases are present, =< 5 x ULN
* Alkaline phosphatase =< 2.0 x ULN; if bone or liver metastases are present, =< 5 x ULN
* Bilirubin =< 1.5 x ULN
* Creatinine =< 1.5 x ULN OR calculated or measured creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine above institutional normal
* Women of childbearing potential must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately

  * Pregnancy testing: women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 or GDC-0449 (serum or urine); a pregnancy test (serum or urine) will be administered every cycle if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of study drug; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing study drug, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097 and GDC-0449
  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
    * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun; if a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Patient must have the ability to understand and the willingness to sign a written informed consent document
* Patients must have a corrected QT (QTc) interval of =< 450 msec in males and a QTc =< 470 msec in females as measured by electrocardiogram (ECG) using Bazett's formula

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (4 weeks for those who received radiation therapy of > 5% of their total marrow volume; 6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from toxicities related to prior therapy are not eligible to participate in this study; patients who have been administered GDC-0449 or RO4929097 as part of a single or limited dosing study, such as a phase 0 study, should not necessarily be excluded from participating in this study solely because of receiving prior GDC-0449 or RO4929097
* Patients may not have received any other investigational agents within the preceding 30 days or five half- lives of the drug and must have full recovery from any acute effects of these investigational therapies
* Patients must not have received prior treatment with either a gamma-secretase or hedgehog inhibitor
* Patients with a requirement for antiarrhythmics or other medications known to prolong QTc
* Patients must not receive any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (i.e. megestrol acetate, bisphosphonates); these medications must have been started 1 month prior to enrollment on this study
* Patients with a prior history of seizures
* Patients with known active brain metastases will be excluded from this clinical trial; patients with prior treated brain metastases (treated and stable for >= 1 month) are allowed, providing that they were not accompanied by seizures and that a baseline brain magnetic resonance imaging (MRI) scan prior to study entry demonstrates no current evidence of progressive brain metastases
* Any patient requiring chronic maintenance of white blood cell counts or granulocyte counts through the use of growth factor support (e.g. Neulasta, Neupogen)
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449 or RO4929097
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients with clinically active liver disease, including active viral or other hepatitis or cirrhosis, are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* GDC is a cytochrome P450 2C9 (CYP2C9) inhibitor; CYP2C9 is an enzyme that metabolizes warfarin sodium (Coumadin) into an inactive metabolite; patients who are on warfarin anticoagulation are allowed to participate as long as they fit the following 4 criteria:

  * They are therapeutic on a stable warfarin dose
  * Their international normalized ratio (INR) target range is no greater than 3
  * They are monitored with weekly INR testing
  * They have no active bleeding or pathological condition that carries high risk of bleeding.
  * Other anticoagulants, including enoxaparin (Lovenox) and fondaparinux (Arixtra) are also permitted
* Caution should be exercised when dosing RO4929097 and GDC-0449 concurrently with CYP2C8, CYP2C9, CYP2C19, and CYP3A4 substrates; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP2C8, CYP2C9, CYP2C19, and CYP3A4 should be switched to alternative medications to minimize any potential risk; investigators will make every effort to switch to another agent and assess the eligibility of the patient to participate in this study
* Baseline QTc > 450 msec in males and QTc > 470 msec in females by ECG using Bazett's formula
* Patients without accessible tumor or who refuse serial biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
MTD and/or RP2D of gamma-secretase/Notch signalling pathway inhibitor RO4929097, determined according to incidence of DLT, graded using the NCI CTCAE | 6 weeks
Occurrence of adverse events and the associated National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade | Up to 30 days after completion of study treatment
Occurrence of DLTs and the associated NCI CTCAE grade | 6 weeks

SECONDARY OUTCOMES:
Change in gene expression levels | Baseline to up to 30 days
  Will be summarized with descriptive statistics appropriate to such distributions.
Change in percentage of select BCSC biomarkers in the Hh and Notch signaling pathways | Baseline to 2 weeks of intervention
  Will be summarized with standard descriptive statistics (N, median, mean, standard deviation, minimum, maximum, and the 90% confidence interval for the mean).
Max concentration (Cmax), time to Cmax (tmax), terminal half-life (t1/2), area under curve 0-infinity (AUC0-inf), AUC 0-next dose (AUCtlast), accumulation index (AI), Cmax steady state (Css, max), and min concentration steady state (Css, min) | Course 1 days 1-3 or days -2, -1, and 1; course 1 days 17 and 21; and course 2 days 1, 7, 10, and 11
  Single and multiple-dose PK parameters summarized with standard descriptive statistics (N, median, mean, standard deviation, minimum, maximum, and the 90% confidence interval for the mean).
Measurement of tumor response using RECIST criteria before and after treatment | Up to 30 days after completion of study treatment
  Will be described by point estimates and exact 90% confidence intervals for proportions using Wilson's method.
Pharmacogenetics (PG) parameters, including, but not limited to, metabolizing enzymes (e.g., CYP3A5, 2C9, and UGT1A1) and transporters (e.g., ABCG2 and ABCB1) | Baseline
  Summarized with standard descriptive statistics (N, median, mean, standard deviation, minimum, maximum, and the 90% confidence interval for the mean).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan